CLINICAL TRIAL: NCT05047068
Title: OCS Heart Perfusion (OHP) Post-Approval Registry
Brief Title: OCS Heart Perfusion Post-Approval Registry
Status: Active, not recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCSHEART-01-ClinPAS
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- OCS DBD Heart Primary Analysis Population: 200 adult primary heart transplant recipients of OCS perfused DBD donor hearts that meet the FDA-approved indication for use except for the following recipient exclusion criteria:
  * Concurrent (multi-organ transplant) or previous solid organ or bone marrow transplant; or
  * On renal dialysis at time of transplant
  Interventions: Device: OCS Heart System
- OCS DCD Heart Primary Analysis Population: 150 adult primary heart transplant recipients of OCS perfused DCD donor hearts that meet the FDA-approved indication for use except for the following recipient exclusion criteria:
  * Concurrent (multi-organ transplant) or previous solid organ or bone marrow transplant; or
  * On renal dialysis at time of transplant
  * Transplanted with DCD heart with warm ischemic time > 30 minutes (warm ischemic time is defined as: Time from when mean systolic blood pressure (SBP) is < 50 mmHg or peripheral saturation < 70% to aortic cross-clamp and administration of cold cardioplegia in the donor).
  Interventions: Device: OCS Heart System
- Other OCS Heart Analysis Population: Any/all other recipients of OCS Heart perfused donor hearts outside of the DBD and DCD indications above will be collected in the respective arm of this registry until the enrollment of the PAP of that arm is completed (200 for DBD and 150 for DCD).
  Interventions: Device: OCS Heart System

INTERVENTIONS:
Device: OCS Heart System — The TransMedics® OCS Heart System is a portable system available for ex-vivo maintenance of a donor heart in a metabolically active and beating state.
  The OCS Heart System's innovative technology was designed to comprehensively overcome the historical limitations of cold storage. The OCS Heart System expands the utilization of donor hearts by enabling the use of donor hearts deemed unsuitable for procurement and transplantation at initial evaluation due to limitations of cold static cardioplegic preservation.

SUMMARY:
The objective of this post-approval registry is to provide additional real-world evidence of the performance of the OCS Heart System to preserve DBD and DCD donor hearts.

DETAILED DESCRIPTION:
Multi-center, observational post-approval registry to:

1. compare patient and graft survival of adult primary heart transplant recipients receiving DBD donor hearts perfused and assessed on the OCS Heart System compared to adult recipients of DBD donor hearts preserved using ischemic cold storage hearts (Control) at the same Registry centers over the same time period, and
2. compare patient and graft survival of adult primary heart transplant recipients receiving DCD donor hearts perfused and assessed on the OCS Heart System compared to adult recipients of DBD donor hearts preserved using ischemic cold storage hearts (Control) at the same Registry centers over the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Adult primary heart transplant recipients of DBD or DCD donor hearts perfused on the OCS Heart System.

Recipient Exclusion Criteria:

* Concurrent (multi-organ transplant) or previous solid organ or bone marrow transplant; or
* On renal dialysis at time of transplant.

Donor Exclusion Criteria (for DCD Donor Hearts only):

* Warm ischemic time > 30 minutes (warm ischemic time is defined as: Time from when mean systolic blood pressure (SBP) is < 50 mmHg or peripheral saturation < 70% to aortic cross-clamp and administration of cold cardioplegia in the donor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult primary heart transplant potential recipients on the waiting list for heart transplantation at the participating Registry centers.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Patient Survival | One year post-heart transplant
  Patient survival at one-year post-heart transplant.

OTHER OUTCOMES:
Safety Endpoint | 6 months post-heart transplant
  Heart graft survival at 6 months post-heart transplant.
Long Term Patient Survival | 5 years post-heart transplant
  K-M Patient survival at 1, 2, 3, 4 and 5 years post-transplant
Long Term Graft Survival | 5 years post-heart transplant
  K-M Graft survival at 6mo, 1, 2, 3, 4 and 5 years post-transplant

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Cedars Sinai, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York
  - Montefiore, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White, Dallas, Texas
  - Medical City Dallas, Dallas, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin